CLINICAL TRIAL: NCT03276026
Title: A Randomized Prospective Study to Compare the Effectiveness of Neostigmine Versus Sugammadex in Length of PACU Stay in ASA II and III Patients Undergoing Sleeve Gastrectomy Bariatric Surgery
Brief Title: A Study to Compare Neostigmine vs Sugammadex in Length of PACU Stay in Patients Undergoing Sleeve Gastrectomy Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left the Institution.
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VirtuaHealth
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Nausea and Vomiting; Respiratory Conditions Due to Other External Agents
Keywords: sugammadex; post anesthesia care unit recovery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group/Neostigmine (Active Comparator): The control group will be the 63 patients who receive Neostigmine in a dose of 5mg, along with the anti-cholinergic glycopyrrolate 0.6mg.
  Interventions: Drug: Neostigmine
- Study Group/Sugammadex (Active Comparator): 63 patients will be given Sugammadex in a dose of 2mg/kg if the train of four twitch count is 2 and 4mg/kg if the twitch response has reached 1-2 post-tetanic counts with no twitch response to train of four.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Sugammadex is used for the reversal of neuromuscular block in surgery that requires deep blockade to facilitate surgical procedures.
  Arms: Study Group/Sugammadex
Drug: Neostigmine — Neostigmine is used for the reversal of neuromuscular block in surgery that requires deep blockade to facilitate surgical procedures.
  Arms: Control Group/Neostigmine

SUMMARY:
The investigators will track bariatric patients who received sugammadex versus neostigmine in the post anesthesia care unit until discharge and assess their length of stay and possible nausea / vomiting / hypoxia episodes.

DETAILED DESCRIPTION:
During their preadmission testing, patients planning to undergo sleeve gastrectomy bariatric surgeries will be consented (by having them sign consent forms) and recruited for the study. A trained individual will track these patients after the surgery in the post anesthesia care unit until discharge and assess their length of stay and possible nausea / vomiting. The exact time the investigators are looking to assess is patient arrival to the post anesthesia care unit until patient ready for discharge when the anesthesiologist writes the anesthesia evaluation. The time the reversal agent is administered during the start of skin closure until patient medically ready to leave the post anesthesia care unit will also be taken into account. Blinded to the treatment group, the trained individual will ask each patient every 15 minutes after arrival to the post anesthesia care unit if they are experiencing nausea or vomiting. As an exploratory measure, the trained individual will assess the patient at these same times (every 15 minutes) and determine their oxygen saturation. The investigators will take all the data from the observations and use statistical means to measure what is significant. A discussion and conclusion will follow. Finally, the principal investigator will submit the study outcomes to an anesthesia journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients having sleeve gastrectomy
* Surgeries performed by a particular surgeon - Dr. Sam Wasser
* Body Mass Index greater than 35
* American Society of Anesthesiologists Score II and III patients

Exclusion Criteria:

* Patients having a different type of bariatric surgery including but not limited to duodenal switch, gastric bypass, hand-assisted laparoscopic sleeve gastrectomy
* Sleeve gastrectomy's performed by other surgeons than Dr. Sam Wasser.
* Pregnancy
* Allergic to sugammadex, Zofran or scopolamine
* Chronic Obstructive Pulmonary Disease or Asthma that is uncontrolled
* American Society of Anesthesiologists Score I, IV, V patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Thaler, DO, Principal Investigator — Virtua Health, Inc.
Locations (1):
- Virtua Memorial Hospital, Mount Holly, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group/Neostigmine: The control group will be the 34 patients who receive Neostigmine in a dose of 5mg, along with the anti-cholinergic glycopyrrolate 0.6mg.
  Neostigmine: Neostigmine is used for the reversal of neuromuscular block in surgery that requires deep blockade to facilitate surgical procedures.
- Study Group/Sugammadex: 33 patients will be given Sugammadex in a dose of 2mg/kg if the train of four twitch count is 2 and 4mg/kg if the twitch response has reached 1-2 post-tetanic counts with no twitch response to train of four.
  Sugammadex: Sugammadex is used for the reversal of neuromuscular block in surgery that requires deep blockade to facilitate surgical procedures.
Period: Overall Study
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex
Started | 35 | 33
Completed | 34 | 33
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 43 [21 to 70] | 42 [22 to 73] | 42 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Post Anesthesia Care Unit Length of Stay
Description: Determine the difference in length of stay in the post anesthesia care unit from patient arrival until ready for post anesthesia care discharge for the American Society of Anesthesiologists Score II and III patients reversed with Sugammadex versus Neostigmine in sleeve gastrectomy surgeries.
Time Frame: Observations will be made during each patient's stay in the post anesthesia care unit (about 120 minutes).
Measure: Mean (Full Range); unit: minutes
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex
Number analyzed (Participants) | 34 | 33
minutes | 121 [47 to 185] | 119 [47 to 248]

2. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: Assess the incidence of Postoperative Nausea and Vomiting in the American Society of Anesthesiologists Score II and III patients reversed with Sugammadex versus Neostigmine at arrival to the post anesthesia care unit and every 15 minutes while in the post anesthesia care unit, with the prediction that there will be a lower incidence of Postoperative Nausea and Vomiting in the Sugammadex group.
Time Frame: Observations will be made during each patient's stay in the post anesthesia care unit (about 120 minutes).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex
Number analyzed (Participants) | 34 | 33
Participants
  Positive for PONV | 14 | 14
  Negative PONV | 20 | 19

3. Secondary Outcome: Incidence of Respiratory Complications
Description: Assess the incidence of respiratory complications postoperatively specifically looking at oxygen saturation at patient arrival to the post anesthesia care unit and every 15 minutes after arrival to the post anesthesia care unit and any intervention necessary.
Time Frame: Observations will be made during each patient's stay in the post anesthesia care unit (about 120 minutes).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex
Number analyzed (Participants) | 34 | 33
Participants
  Positive for Hypoxia | 2 | 0
  Negative for Hypoxia | 32 | 33

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of signing the informed consent until the discharge from the PACU.
Arm/Group | Control Group/Neostigmine | Study Group/Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 1/34 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group/Neostigmine (N=34) | Study Group/Sugammadex (N=33)
Inability to recover spontaneous respirations post surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient did not adequately reverse from Neostigmine. Patient was given Suggamadex to recover. Subject tidal volume went from 150-200 to 500-600 with return of spontanenous respirations.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall submit each publication to the Virtua Clinical Trials Office for review and approval prior to publication or presentation, which approval shall not be unreasonably withheld.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03276026/Prot_SAP_000.pdf